CLINICAL TRIAL: NCT06865677
Title: Phase II Pilot Study of Sacituzumab Govitecan for Relapsed Ovarian, Endometrial, and Cervical Carcinomas
Brief Title: Sacituzumab Govitecan for Relapsed Ovarian, Endometrial, and Cervical Carcinomas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This protocol was terminated prematurely because the prior principal investigator departed the Institute without treating any participants.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Stanley Lipkowitz, MD, PhD, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10002068; 002068-C
Record Dates: First submitted 2025-03-07; First posted 2025-03-10 (Actual); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Platinum Resistant Epithelial Ovarian Carcinoma; Recurrent Epithelial Endometrial Carcinoma; Recurrent Epithelial Cervical Carcinoma
Keywords: TROP2; ADC; Gynecologic Malignancies; Relapsed
MeSH Terms: conditions — Recurrence | interventions — sacituzumab govitecan; Electrocardiography; Tomography, X-Ray Computed; Loperamide; Octreotide; atropine sulfate-diphenoxylate hydrochloride drug combination; Antiemetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 -Treatment with Sacituzumab Govitecan (SG) (Experimental): Treatment with Sacituzumab Govitecan (SG).
  Interventions: Drug: Sacituzumab Govitecan; Diagnostic Test: EKG; Diagnostic Test: Brain MRI; Diagnostic Test: CT scans; Procedure: Tumor biopsy; Drug: Loperamide; Drug: Octreotide; Drug: Diphenoxylate/Atropine; Drug: Antiemetics

INTERVENTIONS:
Drug: Sacituzumab Govitecan — 10mg/kg administered intravenous (IV) infusion on days 1 and 8 of each 21-day cycle.
  Other Names: Trodelvy
Diagnostic Test: EKG — Screening.
  Other Names: Electrocardiogram
Diagnostic Test: Brain MRI — Screening. Baseline/Cycle 1 Day 1 (within 14 (+3) days.
  Other Names: Brain magnetic resonance imaging
Diagnostic Test: CT scans — Screening. Baseline/Cycle 1 Day 1 (within 14 (+3) days. Subsequent cycle 3 every 3 cycles ±7 days for the first year and then every 4 cycles ±7 days until progressive disease or up to 5 years. End of treatment assessments +14 days.
  Other Names: Computed tomography scans
Procedure: Tumor biopsy — Baseline/Cycle 1 Day 1≤10 days. End of treatment assessments +14 days (optional).
  Other Names: Tumor bx
Drug: Loperamide — For diarrhea. 4 mg initially followed by 2 mg with every episode of diarrhea for a maximum of 16 mg daily.
  Other Names: Immodium
Drug: Octreotide — For diarrhea. 100-150 mcg subcutaneous (SC) three times a day if diarrhea persists.
  Other Names: Sandostatin; Bynfezia; Mycapssa
Drug: Diphenoxylate/Atropine — For diarrhea. 20 mg of diphenoxylate/atropine (Lomotil) administered according to package insert guidelines.
  Other Names: Lomotil
Drug: Antiemetics — For vomiting as clinically indicated.

SUMMARY:
Background:

Cancers of the female reproductive organs often come back after treatment. A drug called sacituzumab govitecan (SG) has been approved for use in other types of cancers. Researchers want to see if SG can also help people with ovarian, endometrial, or cervical cancers.

Objective:

To test SG in people with ovarian, endometrial, or cervical cancers.

Eligibility:

People aged 18 years and older with ovarian, endometrial, or cervical cancer. Their cancers must have returned after at least 2 rounds of standard treatments.

Design:

Participants will be screened. They will have a physical exam with blood and urine tests. They will have imaging scans and a test of their heart function. They also will have biopsies to get new tissues samples taken from their tumors.

SG is infused through a tube attached to a needle inserted into a vein in the arm. Treatment will be given in 21-day cycles. Participants will receive SG on days 1 and 8 of each cycle. Each infusion takes 1 to 3 hours.

Participants may receive SG for up to 5 years. They can continue as long as the drug is helping them. Imaging scans and other tests will be repeated throughout the study period.

Participants will have an end-of-treatment visit within 2 weeks and a safety visit about 30 days after they stop treatment. Physical exams, blood tests, and imaging scans may be repeated.

Participants will then be contacted by phone every 6 months for up to 10 years after their first dose of SG.

Sponsoring Institution:

National Cancer Institute...

DETAILED DESCRIPTION:
Background:

* Human trophoblast cell-surface marker (TROP2) is a surface glycoprotein originally identified in human placental tissue and highly expressed in gynecologic malignancies. TROP2 overexpression in ovarian, endometrial, and cervical cancers is linked to tumorigenicity and poor overall survival.
* Sacituzumab govitecan (SG) is an antibody-drug conjugate (ADC) of an Immunoglobulin G (IgG(kappa)1 monoclonal antibody targeting TROP2 with a chemotherapeutic payload of SN-38. SN-38 is an active metabolite of irinotecan and acts as a topoisomerase I inhibitor.
* Preclinical data suggest that SG induces deoxyribonucleic acid (DNA) damage, replication stress, and tumor shrinkage in drug-resistant ovarian, endometrial, and cervical cancer in vitro and in vivo preclinical models.
* Further clinical and translational studies are needed to better understand SGs clinical activity and biology in relapsed gynecologic cancer patients.

Objective:

-To determine the objective response rate (ORR) of sacituzumab govitecan (SG) in participants with recurrent gynecological malignancies, calculated for each individual tumor histology by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

Eligibility:

* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status <= 1
* Histologically documented, recurrent platinum-resistant epithelial ovarian, primary peritoneal, or fallopian tube cancer (referred to as ovarian cancer); recurrent endometrioid or serous endometrial cancer; or recurrent epithelial cervical cancer
* At least two prior systemic therapeutic regimens
* Measurable disease by RECIST v1.1 criteria with lesions that can be safely biopsied
* No prior TROP2-targeting antibody drug conjugates (ADC)

Design:

* This is an open label, non-randomized Phase II pilot study with one Arm.
* SG will be administered intravenously (IV) at 10 mg/kg on Days 1 and 8 each 21-day cycle.
* Tumor assessments will be time-based: every 9 weeks (+/- 1 week) for the first year and every 12 weeks (+/- 1 week) thereafter until disease progression. Pre-treatment biopsies and serial blood samples will be collected for the correlative studies.
* Treatment will be given for a maximum of 5 years or until disease progression or unacceptable toxicities.
* Up to 66 evaluable participants will be enrolled.

ELIGIBILITY:
* INCLUSION CRITERIA:

Cohort 1 (Ovarian Cancer)

* Participants must have histologically or cytologically confirmed recurrent platinum-resistant (defined as less than six months of platinum-free interval) epithelial (i.e., high grade serous, endometrioid, low grade serous, or clear cell) ovarian carcinoma that is refractory to standard treatment.
* Participants with known BReast CAncer gene (BRCA) mutated tumors should have received a poly(ADP-ribose) polymerase (PARP) inhibitor maintenance or treatment.
* Participants without known BRCA mutation and platinum-resistant tumors must have had prior bevacizumab or not eligible for bevacizumab-based therapy (i.e., history of proteinuria).

Cohort 2 (Endometrial Cancer)

* Participants must have histologically or cytologically confirmed recurrent epithelial (i.e., endometrioid or serous) endometrial carcinoma that is refractory to standard treatment.
* Participants must have received prior anti-programmed cell death-1 (PD-1)/programmed death-ligand 1 (PD-L1)-based therapy or not eligible for anti-PD-1/PD-L1-based therapy.

Cohort 3 (Cervical Cancer)

-Participants must have histologically or cytologically confirmed recurrent epithelial cervical (i.e. squamous or adeno) carcinoma that is refractory to standard treatment.

Note: Participants with a history of human papilloma virus infection (i.e., positive human papillomavirus (HPV deoxyribonucleic acid (DNA testing) are eligible.

-Participants must have received prior bevacizumab-based therapy or not eligible for bevacizumab-based therapy (i.e., history of proteinuria).

Note: Platinum chemotherapy administered concurrent with primary radiation (i.e., weekly cisplatin) is not counted as a systemic chemotherapeutic regimen for management of persistent or recurrent carcinoma of the cervix.

All Cohorts

* Participants must have received at least two systemic therapies including at least one platinum-based therapy regimen.
* Participants must have radiographically measurable disease, per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, and safely biopsiable lesion.
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status <= 1
* Adequate organ and marrow function as defined below:

  * Hemoglobin (Hgb) >= 9.0 g/dL
  * Absolute neutrophil count (ANC) >= 1,500/mcL
  * Platelets >= 100,000/mcL
  * White Blood Cell count (WBC) >= 3,000/mcL
  * Total bilirubin <= 1.5 x upper limit of normal (ULN) (<= 3 x ULN in participants with known/suspected Gilbert's disease)
  * Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT) <= 2.5 x ULN
  * Serum creatinine <= 1.5 x ULN or estimated glomerular filtration rate (GFR) >= 30 ml/min/1.73 m^2
* Participants with suspicion or prior history of treated central nervous system (CNS) metastases with no evidence of active disease (assessed by magnetic resonance imaging (MRI) or contrast computed tomography (CT) scan of the brain and spinal column) are eligible if pretreatment brain MRI demonstrate no evidence of disease in the past 4 weeks prior to entry.
* Major surgical procedure, other than for diagnosis, must not occur within 4 weeks prior to the first dose of study treatment. Participants must have recovered adequately from the toxicity and/or complications from the intervention prior to starting the study drug.
* Participants with prior cancer-directed therapy must have a washout period of 3 weeks prior to the first dose of study treatment.
* Participants with prior cancer-directed immunotherapy-based therapy must have a washout period of 4 weeks prior to the first dose of study treatment.
* Human immunodeficiency virus (HIV)-infected participants are eligible if on stable dose of highly active antiretroviral therapy (HAART), a cluster of differentiation 4 (CD4) count >= 200 cells/mcL, and an undetectable viral load (VL).
* Hepatitis B virus (HBV) positive participants are eligible if they have been treated or are on an appropriate course of antivirals at study entry.
* Participants with a history of hepatitis C virus (HCV) infection (i.e., positive HCV antibody test) must have been treated and cured (undetectable HCV VL at screening). Participants with HCV infection who are currently on treatment are eligible if they have an undetectable HCV VL.
* Individuals of child-bearing potential (IOCBP) must agree to use an effective method of contraception (barrier, surgical sterilization, abstinence) prior to study entry, for the duration of study participation, and for at least 6 months after the last dose of study drug.
* IOCBP must undergo pregnancy testing at screening and must not be pregnant in order to take part. Note: In these cases, a negative Beta-human chorionic gonadotropin (Beta-human chorionic gonadotropin (hCG) (urine or blood) is required.
* Nursing participants must discontinue nursing and/or not begin nursing until 1 month after the last dose of study drug.
* Ability of participants to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Participants who are receiving any other investigational agents
* Primary platinum-refractory ovarian cancer (defined as progression while on the upfront platinum-based therapy)
* Participants with any other concomitant invasive malignancies
* History of severe hypersensitivity or allergic reactions attributed to compounds of similar chemical or biologic composition to sacituzumab govitecan (SG), Camptosar; irinotecan; 7-ethyl-10-{4-[1-piperidino]-1-piperidino}carbonyoxycamptothecin (SN-38), or irinotecan.
* Prior treatment with trophoblast cell-surface marker (TROP2)-targeting antibody drug conjugates (ADC). Participants with prior use of other ADCs are eligible.
* Prior treatment with topoisomerase 1 inhibitors i.e., topotecan
* Symptomatic or untreated brain/central nervous system (CNS) metastases
* Participants who require treatment with uridine diphosphate glucuronosyltransferase (UGT1A1) inhibitors.
* Participants with known homozygous UGT1A1*28 allele if tested during the previous treatment.
* Participants with active infection requiring antibiotics.
* Participants who have not recovered from toxicities or adverse events (AE) related to prior therapy to Grade <= 1 with the following exceptions.

  * Participants with platinum related hypomagnesemia (on replacement) are eligible.
  * Participants with auto-immune thyroid dysfunction on stable replacement therapy are eligible.
  * Participants with any grade alopecia or grade 1 or 2 neuropathy are eligible.
* Participants with a history of gastrointestinal (GI) perforation or hemorrhage (> 30mL bleeding/episode) fistula or hemoptysis within 3 months prior to initiation of study therapy, intra-abdominal abscess in the 6 months prior to entry, history of ascites or pleural effusion requiring paracentesis or thoracentesis in the 4 weeks prior to initiation of study therapy or history of bowel obstruction within 3 months prior to initiation of study therapy.
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during SG treatment or within 5 months after the final dose of SG. Note: Seasonal flu vaccines that do not contain a live virus and locally authorized/approved Coronavirus disease 2019 (COVID-19) vaccines are permitted
* Participants with severe uncontrolled intercurrent illness that would limit compliance with study requirements, evaluated by history, physical exam, and chemistry panel.

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2025-06-09 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Conlon, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the National Institutes of Health (NIH) Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the intramural research program (IRP), as of January 25, 2023, that is associated with an investigator-initiated intramural research program (ZIA), with a clinical protocol that undergoes scientific review and/or will involve genomic data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: This study will comply with the National Institutes of Health (NIH) Data Management and Sharing (DMS) Policy. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Data from this study may be requested by contacting the principal investigator (PI). Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_002068-C.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were enrolled in Arm 1/Cohort 1 - Participants with recurrent/metastatic ovarian carcinoma, and Arm 2/Cohort 2 - Participants with recurrent/metastatic endometrial carcinoma.
Groups:
- Arm 1/Cohort 3 -Treatment With Sacituzumab Govitecan (SG); Participants Not Assigned to an Arm/Cohort - Treatment With Sacituzumab Govitecan (SG): Treatment with Sacituzumab Govitecan (SG).
  Sacituzumab Govitecan: 10mg/kg administered intravenous (IV) infusion on days 1 and 8 of each 21-day cycle.
Period: Overall Study
Arm/Group | Arm 1/Cohort 3 -Treatment With Sacituzumab Govitecan (SG) | Participants Not Assigned to an Arm/Cohort - Treatment With Sacituzumab Govitecan (SG)
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — Screen failure | 1 | 0
Not completed — Participant no longer eligible before start of conditioning | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants Not Assigned to an Arm/Cohort - Treatment With Sacituzumab Govitecan (SG) | Arm 1/Cohort 3 -Treatment With Sacituzumab Govitecan (SG) | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 | 65 | 56 (12.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Partial Response or Complete Response) of Sacituzumab Govitecan in Participants With Recurrent Gynecological Malignancies, Calculated for Each Individual Tumor Histology by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: Overall Response Rate (the fraction of Partial Response (PR) or Complete Response (CR) will be calculated along with a 95% confidence interval for each cohort. The proportion of participants who achieve a response will be reported separately for each cohort, along with 95% confidence intervals (Clopper-Pearson). Response was assessed by the RECIST v1.1. Complete Response is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to 22 days.
Population: This endpoint was not done. This protocol was terminated prematurely because the prior principal investigator departed the Institute without treating any participants.
Arm/Group | Arm 1/Cohort 3 -Treatment With Sacituzumab Govitecan (SG) | Participants Not Assigned to an Arm/Cohort - Treatment With Sacituzumab Govitecan (SG)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Median Duration of Response (DOR) of Sacituzumab Govitecan (SG)
Description: Duration of response (DOR) will be calculated by the Kaplan-Meier method, starting at date response was identified until progression or the response is declared to have ended, if the participants have a PR or CR. The median DOR will be reported along with a 95% confidence interval by cohort. Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Complete Response is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Progressive Disease is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The appearance of one or more new lesions is also considered progressions.
Time Frame: Up to 22 days.
Population: as for outcome 1
Arm/Group | Arm 1/Cohort 3 -Treatment With Sacituzumab Govitecan (SG) | Participants Not Assigned to an Arm/Cohort - Treatment With Sacituzumab Govitecan (SG)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Overall Survival of Participants Receiving Sacituzumab Govitecan (SG)
Description: Overall Survival (OS) will be calculated from on-study date until date of 10-year follow-up, using the Kaplan-Meier method by cohort. The ten-year OS rate, which is the percentage of people in a study or treatment group who are alive ten years after their initiation of the study treatment. The median OS will be reported along with a 95% confidence interval by cohort.
Time Frame: Up to 22 days.
Population: as for outcome 1
Arm/Group | Arm 1/Cohort 3 -Treatment With Sacituzumab Govitecan (SG) | Participants Not Assigned to an Arm/Cohort - Treatment With Sacituzumab Govitecan (SG)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Progression Free Survival (PFS) of Participants Receiving Sacituzumab Govitecan (SG)
Description: Progression Free Survival (PFS) will be calculated from on-study date until date of progression or death without progression, using the Kaplan-Meier method by cohort. The median PFS will be reported along with a 95% confidence interval by cohort. Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Progressive Disease is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The appearance of one or more new lesions is also considered progressions.
Time Frame: Up to 22 days.
Population: as for outcome 1
Arm/Group | Arm 1/Cohort 3 -Treatment With Sacituzumab Govitecan (SG) | Participants Not Assigned to an Arm/Cohort - Treatment With Sacituzumab Govitecan (SG)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Adverse Events (AE) Per Common Terminology Criteria for Adverse Events (CTCAE) v5.0, by Type and Grade of Toxicity
Description: Safety will be reported by describing adverse events (AE) per CTCAE v5.0, by type and grade of toxicity. A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned. Grade 1 is mild. Grade 2 is moderate. Grade 3 is severe. Grade 4 is life-threatening. Grade 5 is death related to adverse event.
Time Frame: Up to 22 days.
Population: This protocol was terminated prematurely because the prior principal investigator departed the Institute without treating any participants.
Measure: Number; unit: Adverse events
Arm/Group | Arm 1/Cohort 3 -Treatment With Sacituzumab Govitecan (SG) | Participants Not Assigned to an Arm/Cohort - Treatment With Sacituzumab Govitecan (SG)
Number analyzed (Participants) | 1 | 1
Adverse events | 0 | 0

6. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Up to 22 days.
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1/Cohort 3 -Treatment With Sacituzumab Govitecan (SG) | Participants Not Assigned to an Arm/Cohort - Treatment With Sacituzumab Govitecan (SG)
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality and Adverse Events was monitored/assessed up to 22 days.
Description: This protocol was terminated prematurely because the prior principal investigator departed the Institute without treating any participants.
Arm/Group | Arm 1/Cohort 3 -Treatment With Sacituzumab Govitecan (SG) | Participants Not Assigned to an Arm/Cohort - Treatment With Sacituzumab Govitecan (SG)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-10-24): https://cdn.clinicaltrials.gov/large-docs/77/NCT06865677/Prot_SAP_000.pdf
  • Informed Consent Form (2025-08-12): https://cdn.clinicaltrials.gov/large-docs/77/NCT06865677/ICF_001.pdf